CLINICAL TRIAL: NCT03501537
Title: Soft Tissue Conditioning to for the Treatment of Peri-implantitis in the Lack of Keratinised Mucosa
Brief Title: Association of Keratinised Mucosa Around Implants and Teeth With Peri-implant/Periodontal Disease and Soft Tissue Conditioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18002909C
Record Dates: First submitted 2018-04-04; First posted 2018-04-18 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Peri-Implantitis; Soft Tissue; Bone Gain
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Single-prospective one-arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical treatment with free gingival graft (Experimental): Free gingival graft harvested from the palate will be placed around the diseased implant
  Interventions: Procedure: Free gingival graft obtained from the palate and debridement of the peri-implant lesion

INTERVENTIONS:
Procedure: Free gingival graft obtained from the palate and debridement of the peri-implant lesion — granulation tissue debridement and grafting of a free gingival strip obtained from the palate

SUMMARY:
Lack of keratinised mucosa around dental implants and teeth is associated with plaque accumulation and worse tissue conditions. However, there is lack of data on the influence of the presence/lack of keratinised mucosa on the periodontal condition. Hence, soft tissue conditioning by grafting with a gingival graft is aimed at improving the quality of the peri-implant conditions

ELIGIBILITY:
Inclusion Criteria:

* Partial edentulous patients with adjacent teeth
* Lack of keratinised mucosa
* Healthy patient

Exclusion Criteria:

* Pregnancy
* Complete edentulous patients
* Patients taking any medication
* Smokers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Peri-implant conditions | 12 months after implant loading
  Probing pocket depth measured in mm, bleeding on probing recorded as yes/no (I/0), suppuration as recorded as yes/no (I/0)

SECONDARY OUTCOMES:
Association of keratinised mucosa/gingiva with periodontal and peri-implant conditions | 12 months after implant loading
  keratinised mucosa (mm) and keratinised gingiva (mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Implantologia Cirugia Oral y Maxilofacial, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Parpaiola A, Cecchinato D, Toia M, Bressan E, Speroni S, Lindhe J. Dimensions of the healthy gingiva and peri-implant mucosa. Clin Oral Implants Res. 2015 Jun;26(6):657-62. doi: 10.1111/clr.12359. Epub 2014 Feb 26. PMID 24611985
- [Derived] Monje A, Blasi G. Significance of keratinized mucosa/gingiva on peri-implant and adjacent periodontal conditions in erratic maintenance compliers. J Periodontol. 2019 May;90(5):445-453. doi: 10.1002/JPER.18-0471. Epub 2018 Dec 7. PMID 30461016